CLINICAL TRIAL: NCT03588741
Title: Evaluation of Safety Following Immune Tolerance Induction Treatment With Turoctocog Alfa in Patients With Haemophilia A Following Inhibitor Development in NN7170-4213 Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was terminated as the participant withdrew from the trial.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7170-4345; U1111-1187-7323 (Other: WHO); 2016-003821-40 (EudraCT Number)
Record Dates: First submitted 2018-06-12; First posted 2018-07-17 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Turoctocog alfa (Experimental)
  Interventions: Drug: Turoctocog alfa

INTERVENTIONS:
Drug: Turoctocog alfa — Intravenous (i.v., under the skin) administration.A maximum dose of 200 IU/kg daily.
  The maximum treatment period for this trial is 24 months and the patient(s) will be called for visit to the clinic every 3rd month.

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of the trial is to evaluate safety of immune tolerance induction (ITI) treatment with turoctocog alfa (a recombinant factor VIII) in patients who have developed neutralising antibodies against factor VIII after exposure to subcutaneous turoctocog alfa pegol during participation in NN7170-4213 (NCT02994407)

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the NN7170-4213 trial (male, age at least 18 years (part A) and age at least 12 years (part B))
* Development of a confirmed high titre neutralising antibody towards factor VIII (greater than 5 Bethesda Unit) after exposure to subcutaneous turoctocog alfa pegol in the NN7170-4213 trial or development of a confirmed clinically relevant low titre inhibitor (at least 0.6 to below or equal to 5 Bethesda Unit), defined as factor VIII activity measures (recovery) and/or bleedpattern indicating a lack of clinical response to factor VIII treatment

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products, defined as allergic reactions
* Participation in another clinical trial within 1 month before screening (except participation in NN7170-4213)
* Any disorder, except for conditions associated with Haemophilia A which in the investigator's opinion might jeopardise patients' safety or compliance with the protocol
* Currently receiving immune tolerance induction treatment with a factor VIII containing product other than turoctocog alfa

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (13):
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Novo Nordisk Investigational Site, Nantes, France
- Germany (3):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Homburg
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Novo Nordisk Investigational Site, Bornova-IZMIR, Turkey (Türkiye)
- United Kingdom (3):
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 1 trial site in Germany.
Pre-assignment Details: Previously treated participants with severe haemophilia A (FVIII activity <1% according to medical records) who had developed clinically relevant FVIII inhibitors in trial NN7170-4213 were offered immune tolerance induction (ITI) treatment with turoctocog alfa.
Groups:
- Turoctocog Alfa: The participant received intravenous (i.v.) injection of 65 international units per kilogram (IU/kg) turoctocog alfa 3 times per week. The planned treatment duration was for at least 12 months and up to a maximum period of 24 months.
Period: Overall Study
Arm/Group | Turoctocog Alfa
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised of the participant(s) who initiated ITI treatment with turoctocog alfa.
Arm/Group | Turoctocog Alfa
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment.
Time Frame: Month 0 - up to month 12
Population: Safety analysis set (SAS) comprised of the participant(s) who initiated ITI treatment with turoctocog alfa.
Measure: Number; unit: Adverse events
Arm/Group | Turoctocog Alfa
Number analyzed (Participants) | 1
Adverse events | 6

2. Secondary Outcome: Response to FVIII ITI Treatment (Success, Partial Success, Failure, Other)
Description: ITI treatment response was categorized as: 1. Success: Undetectable inhibitor titre <0.6 bethesda units (BU) (or lower limit of quantification [LLoQ] if above 0.6 BU); Normalised FVIII in vivo recovery, defined as ≥0.013 international units (IU) per milliliter per IU per kilogram ((IU/ml)/(IU/kg)) (66% of expected incremental recovery); turoctocog alfa half-life ≥7 hours (based on FVIII activity) after 72 hours treatment-free washout period. 2. Partial success: Inhibitor titre ≤5 BU; Clinical effect of turoctocog alfa therapy as judged by the investigator. 3. Failure (one criterion had to be fulfilled): Failure to attain defined success or partial success after 24 months of ITI treatment with turoctocog alfa; Decrease in inhibitor titre after 12 months of ITI treatment <20% compared to peak titre. 4. Other: Participants not fulfilling the above criteria e.g. early withdrawal from ITI treatment, lack of adherence to recommended ITI protocol etc.
Time Frame: Month 12
Population: FAS comprised of the participant(s) who initiated ITI treatment with turoctocog alfa.
Measure: Count of Participants; unit: Participants
Arm/Group | Turoctocog Alfa
Number analyzed (Participants) | 1
Participants
  Success | 0
  Partial success | 0
  Failure | 0
  Other | 1

ADVERSE EVENTS:
Time Frame: Month 0 - up to month 12
Description: Results are based on the safety analysis set (SAS), which comprised the participant(s) who initiated ITI treatment with turoctocog alfa.
Arm/Group | Turoctocog Alfa
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Turoctocog Alfa (N=1)
Nasopharyngitis (Infections and infestations) | 1 (3)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated as the participant withdrew from the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03588741/Prot_SAP_000.pdf